CLINICAL TRIAL: NCT04794595
Title: Clinical Features and Outcomes of Continuous Blood Purification Versus Non-continuous Blood Purification in Pediatric Patients With Sepsis or Septic Shock
Brief Title: Clinical Features and Outcomes of CBP Versus Non-CBP in Septic Children
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-08
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Children, Only
Keywords: Continuous renal replacement therapy; sepsis; timing
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the volume of 2ml whole blood was stored in EDTA tube
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group with CBP: The child with sepsis should be treated with CBP， but could not receive this treatment for various reasons
  Interventions: Procedure: CBP
- sepsis group without CBP: The child with sepsis should be treated with CBP and received this treatment

INTERVENTIONS:
Procedure: CBP — continuous blood purification can prevent or treat fluid overload in children with septic shock or other sepsis-associated organ dysfunction who are unresponsive to fluid restriction and diuretic therapy management of septic AKI patients, particularly those with hemodynamic instability or fluid overload. Also, it can remove cytokines
  Other Names: traditional therapy
  Groups: sepsis group with CBP

SUMMARY:
The effect of continuous blood purification (CBP) in children is unclear. Also, the timing of early application is still being explored. In this study, we need to explore the efficacy and the timing of application of CBP in children with sepsis or septic shock.

DETAILED DESCRIPTION:
Early intervention of CBP can remove inflammatory factors in patients with sepsis and reduce the damage of inflammatory factors to organs; at the same time, it can also promote the body's immune response, significantly improve immune dysfunction, and restore the body's immune balance. However, the timing of early application of CBP in childhood sepsis is still unclear. Therefore, it is necessary to further explore the treatment and prognosis of this technology in the early treatment of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age of 29d to 18 years old;
* Children diagnosed with sepsis requiring blood purification.

Exclusion Criteria:

* with a history of a duration of PICU stay <24 h
* active bleeding, including cerebral hemorrhage

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with sepsis requiring blood purification to prevent or treat fluid overload or to clear cytokines
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
survival rate | 28 days after hospital discharge
  The survival rate of children in 28 days after hospital discharge

SECONDARY OUTCOMES:
The creatinine level of non-survival children with sepsis | 28 days after hospital discharge
  The creatinine level of non-survival children with sepsis in 28 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lu guoing, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children'S Hospital of Fudan University, Shanghai, Shanghai Municipality, China